CLINICAL TRIAL: NCT01684566
Title: A Multicenter, Open-label, Parallel Group Investigation to Compare the Performance of Standard Of Care (SOC) and Episil® in Combination Versus SOC Alone on Oral Mucositis in Patients Receiving Conditioning Treatment for Hematopoietic Stem Cell Transplantation
Brief Title: A Comparative Investigation of Standard Of Care (SOC) and Episil® in Combination Versus SOC Alone on Oral Mucositis
Acronym: episil(R)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-10-396
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-11

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-Of-Care + episil(R) (Experimental): Standard-Of-Care plus episil® administered as three consecutive pump-strokes for a total volume of 0.45 mL applied 3 times daily and additionally, as needed
  Interventions: Device: episil(R); Other: Oral hygiene procedures
- Standard-Of-Care (Other): Oral hygiene procedures
  Interventions: Other: Oral hygiene procedures

INTERVENTIONS:
Device: episil(R) — episil® is a lipid-based liquid that spreads onto mucosal surfaces and transforms into a protective, strongly bioadhesive FluidCrystal® film after intraoral administration.
  Arms: Standard-Of-Care + episil(R)
Other: Oral hygiene procedures — Oral hygiene by using toothbrush, toothpaste, lip balm and dental floss (if available)

SUMMARY:
To compare the performance of standard of care (SOC) + episil® versus SOC alone on oral mucositis in patients receiving conditioning treatment for hematopoietic stem cell transplantation (HSCT). The primary variable will be the area under the curve (AUC) of oral mucositis scores defined by the World Health Organisation (WHO) oral toxicity scale assessed daily by the investigator over the 28-day study period.

DETAILED DESCRIPTION:
This was multicentre, open-label, randomised parallel-group study. Patients were randomised to one of two parallel treatment groups: episil® in combination with SOC or SOC alone.

The study was originally planned to be conducted in several sites in the following countries: Denmark, Israel, Poland, and Sweden. Following a country-specific Amendment on 20-Feb-2013 and a German Ethical Committee (EC) approval in 07-May-2013, Germany was added to the list of countries where the study would be conducted. No study sites were initiated in Denmark.

The study design was aimed to facilitate direct comparison of the performance of SOC + episil® versus SOC alone. The study was conducted in an open-label manner that is common in trials involving cancer patients, as this takes into the account the ethical issues involved in this indication and patient population. To reduce the likelihood of bias, assignment to study treatment was randomised.

SOC as control group is appropriate and widely used, especially in trials involving cancer patients. In this particular study, basic oral hygiene consisting of brushing, flossing, rinsing and moisturising was taken as the SOC used as control group.

.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age.
2. Has a confirmed diagnosis for which he/she is scheduled for hematopoietic stem cell transplantation (HSCT) of either type of transplant (autologous or allogeneic).
3. Is due to undergo treatment with myeloablative conditioning (radiation-based or non radiation based) before HSCT.

Exclusion Criteria:

1. Will undergo reduced intensity conditioning before HSCT.
2. Has got known allergy to any ingredient in the study product or to peanuts, peppermint oil, or soya.
3. Is pregnant or breast feeding.
4. Has any other concurrent medical condition that, in the opinion of the investigator, would increase the risk to the patient, compromise evaluation of the investigational device, or interfere with the conduct of the study.
5. Has an unstable condition (eg, a psychiatric disorder, a recent history of substance abuse) or is otherwise thought to be unreliable or incapable of complying with the study requirements.
6. Is undergoing treatment with parenteral opioids at enrolment.
7. Uses treatments that promote mucosal healing (eg, palifermin).
8. Uses electrolyte mouthwashes (eg, Caphosol®) or other topical oral treatments (eg, Tantum Verde® (benzydamine), Gelclair®, Fungicidin (nystatin)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Garming-Legert, DDS, PhD., Principal Investigator — Karolinska Institutet
Locations (12):
- Germany (2):
  - Med Klinik und Poliklinik I Universitatsklinikum Carl Gustav Carus, Dresden
  - Abteilung fur Hamatologie und Onkologie Universitatsmedizin an der Georg-August-Universitat, Göttingen
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Centre, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Tel-Aviv Sourasky Medical Centre, Tel Aviv
- Poland (3):
  - Military Institute of Medicine Internal diseases and Haemtalogy Clinic, Warsaw
  - Institute of Haematology and Transfusion Medicine, Warsaw
  - Oncology Center Institute named Maria Sklodowska-Curie Lymph System Cancer Clinic, Warsaw
- Sweden (3):
  - Karin Garming-Legert, Stockholm, Huddinge
  - Lund University Hospital, Lund
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Started | 60 | 56
Treated (ITT) | 57 | 52
Completed | 44 | 49
Not Completed | 16 | 7

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care | Total
Number analyzed (Participants) | 57 | 52 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (15.21) | 49.0 (14.82) | 47.6 (15.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 15 | 42
  Male | 30 | 37 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 56 | 51 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Sweden | 11 | 9 | 20
  Israel | 23 | 23 | 46
  Poland | 13 | 13 | 26
  Germany | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: WHO (World Health Organisation) Oral Mucositis Severity Score During 28 Days of Treatment, Intention to Treat Population
Description: Summary of WHO (World Health Organisation) Oral Toxicity Scores Area under the curve (AUC) over the 28-Day Period ITT Populations.
  A higher score represents a more severe oral mucositis Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: Intention to treat (ITT) and Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 57 | 52
score | 0.63 (0.702) | 0.56 (0.589)

2. Secondary Outcome: Occurrence of Oral Mucositis
Description: Occurrence of oral mucositis (ie, oral mucositis defined as WHO (World Health Organization) oral toxicity scale grade 0-4.
  A higher score represents a more severe oral mucositis Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 57 | 52
participants | 44 | 40

3. Secondary Outcome: Duration of Oral Mucositis, Intention to Treat Population
Description: Duration of oral mucositis during the treatment period of 28 Days. Oral mucositis was graded according to WHO 5 Point grading scale on a daily basis.
  Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: ITT (Intention to treat). There were13 patients in the episil +SOC group and 12 patients in the SOC group who had no data for duration of oral mucositis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 44 | 40
Days | 9.5 (6.85) | 10.7 (6.03)

4. Secondary Outcome: Oral Mucositis Daily Questionnaire (OMDQ)
Description: OMDQ (Oral Mucositis Daily Questionnaire) scale was used to measure Overall Mouth and Throat Soreness This was scored from 0=no soreness to 10=worst possible soreness.
Time Frame: 28 days
Population: Intention to treat(ITT) OMDQ AUC over time. Not all patients reported data from OMDQ therefore there is lower number of patients in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 41 | 36
units on a scale | 2.59 (1.619) | 2.64 (1.539)

5. Secondary Outcome: Oral Mucositis Assessment Scale (OMAS)
Description: Summary of Oral Mucositis Assessment Scale (OMAS) Ulceration and Erythema Scores Extent of ulceration (grade 0-3) and severity of erythema (grade 0-2) according to the OMAS (Oral Mucositis Assessment Scale) assessed by a dental practitioner twice-weekly over the 28-day study period.
  The extent of ulceration was rated as follows:
  0 no lesion
  1. 1 cm2
  2. 1-3 cm2
  3. >3 cm2
  The severity of erythema was assessed as follows:
  0 none
  1. not severe
  2. severe
Time Frame: 28 days
Population: Intention to treat (ITT) Ulceration and Erythema.OMAS was only performed in sites were a dentist was available therefore lower numbers in the analysis.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 23 | 25
score
  Ulceration | 0 (0.21) | 0 (0.20)
  Erythema | 0.3 (0.70) | 0.5 (1.39)

6. Secondary Outcome: Hospital Stay, Days
Description: Duration of hospital stay (time from admission to discharge)
Time Frame: 28 days
Population: Intention to treat (ITT) Hospital stay, days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 57 | 52
Days | 23.7 (4.45) | 24.5 (3.43)

7. Primary Outcome: WHO (World Health Organisation) Oral Mucositis Severity Score During 28 Days of Treatment, Per Protocol Population
Description: Summary of WHO (World Health Organisation) Oral Toxicity Scores AUC Over the 28-Day Period Per protocol population.
  A higher score represents a more severe oral mucositis Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: Per Protocol (PP) without Last observation carried over(LOCF)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 37 | 49
score | 0.39 (0.402) | 0.56 (0.587)

8. Secondary Outcome: Occurence of Oral Mucositis, Per Protocol Population
Description: Occurrence of oral mucositis (ie, oral mucositis defined as WHO (World Health Organisation) oral toxicity scale grade 0-4
  A higher score represents a more severe oral mucositis Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: Per Protocol (PP)
Measure: Number; unit: participants
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 37 | 49
participants | 28 | 37

9. Secondary Outcome: Duration of Oral Mucositis, Per Protocol Population
Description: Duration of oral mucositis during the treatment period of 28 Days. Oral mucositis is graded according to the 5-point oral mucositis WHO scale Grade 0 No mucositis Grade 1 Soreness ± erythema, no ulceration Grade 2 Erythema, ulcers. Patients can swallow solid diet Grade 3 Ulcers, extensive erythema. Patients cannot swallow solid diet Grade 4 Oral mucositis to the extent that alimentation is not possible
Time Frame: 28 days
Population: Per Protocol (PP). There were 9 patients in the episil +SOC group and 12 patients in the SOC group who had no data for duration of oral mucositis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Number analyzed (Participants) | 28 | 37
Days | 7.4 (5.85) | 10.1 (5.58)

ADVERSE EVENTS:
Time Frame: Adverse event was collected during the treatment period day 1-28 +follow-up 14 Days +/- 2 Days after last application
Arm/Group | Standard-Of-Care + Episil(R) | Standard-Of-Care
Serious Adverse Events (participants affected / at risk) | 4/57 | 1/52
Other Adverse Events (participants affected / at risk) | 26/57 | 23/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-Of-Care + Episil(R) (N=57) | Standard-Of-Care (N=52)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pulmonay haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-Of-Care + Episil(R) (N=57) | Standard-Of-Care (N=52)
Vomiting (Gastrointestinal disorders) | 10 (10) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 6 (6)
febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 9 (9)
Pyrexia (General disorders) | 8 (8) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days